CLINICAL TRIAL: NCT03140696
Title: Formative Research on the Use of Egg as a Nutritional Supplement for Young Bangladeshi Children and Breast Milk Nutrient Content of Bangladeshi Women
Brief Title: Formative Research Study to Address Protein Intake in Children and Analysis of Breast Milk Nutrient Content in Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PR-16094
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-01

CONDITIONS: Protein Malnutrition
MeSH Terms: conditions — Kwashiorkor | interventions — Eggs; Milk, Human

STUDY DESIGN:
Intervention Model Description: The children will be randomly allocated to one of the three types of food (egg alone or egg + RUSF or egg + breast milk) in a crossover design.
  Each of the diets (egg alone or egg + RUSF or egg + breast milk) will be offered for 2 days each. The order of diets will be randomly allocated over a period of 6 days. There would be 6 possible permutations and combinations of the order of the diets over this 6 days sequential period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chicken egg alone (Experimental): A chicken egg alone will be offered for 2 days by mouth for once a day
  Interventions: Dietary Supplement: Egg Alone
- Egg and RUSF (Experimental): A chicken egg and Ready to use supplementary food (RUSF) will be offered for 2 days by mouth for once a day
  Interventions: Dietary Supplement: Egg and ready to use supplementary food (RUSF)
- Egg and breast milk (Experimental): A chicken egg and Mother's breast milk will be offered for 2 days by mouth for once a day
  Interventions: Dietary Supplement: Egg and breast milk

INTERVENTIONS:
Dietary Supplement: Egg Alone — A chicken egg will be offered for 2 days
  Arms: Chicken egg alone
Dietary Supplement: Egg and ready to use supplementary food (RUSF) — A chicken egg and ready to use supplementary food (RUSF) will be offered for 2 days
  Arms: Egg and RUSF
Dietary Supplement: Egg and breast milk — A chicken egg and breast milk will be offered for 2 days
  Arms: Egg and breast milk

SUMMARY:
This formative research seeks to explore the use of egg (as a potential source of protein) as nutritional supplement for young children aged 6-8 months of either sex and breast milk composition of mothers of infants under 6 months old living in an urban slum of Dhaka city, Bangladesh.

DETAILED DESCRIPTION:
Inadequate dietary protein intake and prolonged undernourishment can lead to short term and long-term consequences, which can deplete financial, physical, and social capital, further exacerbating the cycle of undernutrition. Subsequently, undernutrition contributes to the difficulty in achieving sustainable development and alleviating people from poverty. Children are a particular focus of interest because of the formative impact that nutrition can have on development. This is particularly relevant for the 159 million children from low and middle-income countries (LMICs) who are already stunted and many more are at risk of stunting. Understanding how to prevent child undernutrition is imperative to the future development of these children from LMICs. There is no study done so far to understand the quantity, preference and quality of egg protein intake in young children living in LMICs with high burden of undernutrition. In this context, eggs can serve as a potential source of protein to meet the unmet need of protein especially children living in resource-poor environments. Eggs contain high concentrations of choline - an important precursor of phospholipids, which can prevent adverse pregnancy outcomes, neural tube defects, changes in brain structure and function in offspring, and impaired language development during early childhood. Evidence is limited on the support of egg-related interventions for better nutrition outcomes in children from developing countries. Also there is very little evidence on the association between mother's breast milk composition with child's nutritional status.

ELIGIBILITY:
Inclusion Criteria:

(i) consuming complementary food (liquid or semi-solid or solid food) other than breast milk at least once daily; (ii) free from any acute or chronic illness (es); (iii) no known case of congenital abnormality or chromosomal disorder, and (iii) no history of micro-nutrient or food supplementation in last two weeks prior to enrollment (iv) should be breastfed but not exclusively breastfed

Exclusion Criteria:

* Children whose parents/caregivers refuse to provide informed consent will not be enrolled

Ages: 6 Months to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Ideal mode of feeding egg to young infants 6-8 months of age | 2 days
  Each of the diets (egg alone or egg + RUSF or egg + breast milk) will be offered for 2 days each. The order of diets will be randomly allocated over a period of 6 days.On the first day, the child will be acclimatized with the given regime, and on second day, the mother will be asked to rate the offered food by using a 7-point Hedonic Scale in terms of colour, flavour, appearance and overall liking. A fixed amount of food will be offered. The food offered would be weighed before consumption and the left over will also be weighed to measure the actual amount of food consumed by the children. Total amount of offered food taken by the children will also be recorded. During the feeding time, field research assistants will observe the feeding session by using a structured tool. This combined approach (Hedonic scale and amount of food taken) will be used to determine the ideal mode of feeding of an egg by young infants.

CONTACTS AND LOCATIONS:
Overall Officials: Muttaquina Hossain, MPH, Principal Investigator — Research Investigator
Locations (1):
- icddr,b Mirpur Field site, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
The data will be entirely a property of organization and will be under lock and key under Principal Investigator. No participant data will make available to public without participants concents